CLINICAL TRIAL: NCT05801939
Title: Phase 2 Study of Cevostamab Consolidation Following BCMA CAR T Cell Therapy for Relapsed/Refractory Multiple Myeloma
Brief Title: Cevostamab Following CAR T Cell Therapy for RRMM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 853124, UPCC 02423
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cevostamab (Experimental)
  Interventions: Drug: Cevostamab

INTERVENTIONS:
Drug: Cevostamab — Cevostamab will be given as an IV infusion once every 3 weeks, starting roughly 10 weeks (day 70 +/- 4 days) post-CAR T cell infusion, with subjects planned to receive 8 cycles initially. Subjects receive a single step-up dose of 3.6 mg of cevostamab on cycle 1, day 1 (C1D1), followed by the recommended target dose (160 mg, 132mg, or 90 mg based on results of safety run-in data and safety review) on C1D8. Myeloma responses are assessed every cycle, and a repeat bone marrow aspirate and biopsy (BMbx) is performed at the start of cycle 8. If participants are not in an MRD-negative CR at this timepoint (or if the BM bx is inevaluable/indeterminate for CR or MRD testing), they continue with another 8 cycles (C9-16) of cevostamab. If they are in MRD-negative CR at start of C8, they stop therapy after receiving this cycle and are observed.

SUMMARY:
This is a Phase 2, open-label, single-arm, single stage, single-institution study, with an initial safety run-in period. Potential participants with relapsed/refractory myeloma who are undergoing standard of care, commercially-available BCMA-directed CAR T cell therapy may be identified pre-CAR T cell infusion but are not consented and enrolled until at least 4-6 weeks after CAR T cell infusion, once recovered from acute toxicities. Note: the lymphodepleting chemotherapy and CAR T cell therapy is being administered as part of standard clinical practice and is not considered part of this protocol. Alternative lymphodepleting regimens other than fludarabine and cyclophosphamide (eg in the setting of fludarabine shortages) are acceptable. Cevostamab will be given as an IV infusion once every 3 weeks, starting roughly 10 weeks (day 70 +/- 4 days) post-CAR T cell infusion, with subjects planned to receive 8 cycles initially. Aiming to assess the impact of cevostamab consolidation post-BCMA CAR T cell therapy on rate of MRD-negative complete remission (CR) at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form(s)
2. Age ≥18 years at time of signing Informed Consent Form
3. Ability to comply with the study protocol
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
5. Life expectancy of at least 12 weeks
6. Participants must have relapsed and/or refractory multiple myeloma with therapy that must include a proteasome inhibitor, immunomodulatory drug (IMiD), and anti-CD38 antibody, and have received a BCMA-directed CAR T cell product as standard of care (i.e. not on a clinical trial) as per the current FDA label, between 6 and 10 weeks prior to enrollment, and have not had progressive disease by IMWG criteria since CAR T cell infusion. Patients who have received out-of-specification CAR T cell products are not eligible.

   1. For patients who received ide-cel, they must have had at least 2 prior lines of therapy prior to ide-cel
   2. For patients who received cilta-cel, they must have had at least 2 prior lines prior to cilta-cel, or 1 prior line and be refractory or intolerant to lenalidomide.
7. Agreement to provide bone marrow biopsy and aspirate samples
8. Non-hematologic adverse events from prior anti-cancer therapy resolved to Grade ≤ 1, with the certain exceptions.
9. Measurable disease is not required for study entry
10. Laboratory values as specified in the protocol.
11. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, as defined in the protocol.
12. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined in the protocol.

Exclusion Criteria:

1. Inability to comply with protocol-mandated hospitalization and activities restrictions
2. Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the last dose of study drug

   a. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study drug.
3. Participants who had ≥ Grade 3 cytokine release syndrome (CRS) or immune effector cell-associated neurotoxicity syndrome (ICANS) by ASTCT criteria, or any grade macrophage activation syndrome/hemophagocytic lymphohistiocytosis (MAS/HLH)after CAR-T therapy are excluded
4. Participants who had any grade movement and/or neurocognitive disorder attributed to CAR T cells are excluded.
5. Prior treatment with systemic immunotherapeutic agents, including, but not limited to, cytokine therapy and anti-CTLA4, anti-PD-1, and anti-PD-L1 therapeutic antibodies, within 12 weeks or 5 half-lives of the drug, whichever is shorter, before first cevostamab infusion
6. Known treatment-related, immune-mediated adverse events associated with prior immunotherapeutic agents as specified in the protocol.
7. Treatment with any chemotherapeutic agent, or any other anti-cancer agent (investigational or otherwise) during the time period between CAR T cell infusion and first cevostamab infusion, with certain exceptions.
8. Received systemic immunosuppressive medications (including, but not limited to, steroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, tocilizumab, siltuximab, anakinra, ruxolitinib, and anti-tumor necrosis factor agents), with the exception of corticosteroid treatment ≤ 10 mg/day prednisone or equivalent, within 2 weeks prior to first dose of cevostamab

   a. Participants who received acute, low-dose, systemic immunosuppressant medications (e.g., single dose of dexamethasone for nausea) may be enrolled in the study.

   i. The use of inhaled corticosteroids is permitted. ii. The use of mineralocorticoids for management of orthostatic hypotension is permitted.

   iii. The use of physiologic doses of corticosteroids for management of adrenal insufficiency is permitted.
9. Autologous stem cell transplantation (SCT) within 100 days prior to first cevostamab infusion
10. Prior allogeneic SCT within 12 months prior to first cevostamab infusion. Participants with prior allogeneic SCT must have no evidence for active graft-versus-host-disease (GVHD) and be off all therapy for GVHD for at least 3 months prior to first cevostamab infusion.
11. Prior solid organ transplantation
12. History of autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

    1. Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
    2. Participants with history of immune thromobocytopenic purpura (ITP), autoimmune hemolytic anemia, or other immune-mediated conditions that solely affect blood counts, as long as these conditions are not active at the time of enrollment and subjects otherwise meet hematologic parameters for eligibility, may be eligible with approval from Sponsor Medical Director.
13. Participants with history of confirmed progressive multifocal leukoencephalopathy
14. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
15. History of other malignancy that could affect compliance with the protocol or interpretation of results

    1. Participants with a history of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix are allowed.
    2. Participants with a malignancy that has been treated with curative intent will also be allowed if the malignancy has been in remission prior to first cevostamab infusion.
16. Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, neurodegenerative disease, or CNS involvement by MM

    1. Participants with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 2 years and have no residual neurologic deficits as judged by the investigator are allowed.
    2. Participants with a history of epilepsy who have had no seizures in the past 2 years while not receiving any anti-epileptic medications are allowed.
17. Significant cardiovascular disease (such as, but not limited to, New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, uncontrolled arrhythmias, or unstable angina) that may limit a subject's ability to adequately tolerate a cytokine release syndrome (CRS) event
18. Symptomatic active pulmonary disease or requiring supplemental oxygen
19. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics within 14 days prior to first cevostamab infusion. Empiric or prophylactic antibiotics administered during neutropenia or neutropenic fever without microbiologic evidence of infection do not exclude subjects.

    a. Participants with asymptomatic CMV reactivation (i.e. positive CMV PCR) found at screening may enroll after discussion with the Medical Director.
20. Known or suspected chronic active Epstein-Barr virus (EBV) infection.
21. Recent major surgery within 4 weeks prior to first cevostamab infusion
22. Positive serologic or polymerase chain reaction (PCR) test results for acute or chronic hepatitis B virus (HBV) infection

    a. Participants whose HBV infection status cannot be determined by serologic test results must be negative for HBV by PCR to be eligible for study participation.
23. Acute or chronic hepatitis C virus (HCV) infection

    a. Participants who are positive for HCV antibody must be negative for HCV by PCR to be eligible for study participation.
24. Known history of HIV seropositivity
25. Administration of a live, attenuated vaccine within 4 weeks before first cevostamab infusion or anticipation that such a live attenuated vaccine will be required during the study.
26. Any medical condition or abnormality in clinical laboratory tests that, in the Medical Director's judgment, precludes the subject's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
MRD-negative complete remission (CR) | 12 months
  The proportion of participants who achieve CR as well as MRD-negativity at 12 months post-CAR T cell therapy.

SECONDARY OUTCOMES:
Safety and tolerability (Incidence of Treatment-Emergent Adverse Events) of cevostamab administration post-BCMA CAR T cell therapy | infusion start Day 56 through 30 days post final infusion
  Assessed as the frequency of adverse and serious adverse events, including CRS and neurotoxicity, and frequency of dose reductions and delays.
Feasibility of cevostamab administration post-BCMA CAR T cell therapy | Day 56 and completion through day 203
  Frequency of enrolled subjects who are able to start cevostamab by day 56 post-CAR T cell therapy, and the frequency who complete the 8 planned consolidation doses.
Impact of cevostamab consolidation post-BCMA CAR T cell therapy on other clinical outcomes | 6 and 12 months post-CAR T cell therapy
  Efficacy as assessed by rates of best overall response, partial response (PR), very good partial response (VGPR), complete response (CR), stringent CR (sCR), MRD-negativity

CONTACTS AND LOCATIONS:
Overall Officials: Adam D Cohen, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No